CLINICAL TRIAL: NCT01499043
Title: A Pilot Study of PLX3397 in Advanced Castration-Resistant Prostate Cancer (CRPC) Patients With Bone Metastasis and High Circulating Tumor Cell (CTC) Counts
Brief Title: Pilot Study of PLX3397 in Patients With Advanced Castration-Resistant Prostate Cancer (CRPC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision.
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX108-06
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
Keywords: CRPC; Prostate Cancer; Bone metastasis; Advanced Castration-Resistant Prostate Cancer (CRPC)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pexidartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PLX3397 (Experimental): Participants will take daily oral dose of PLX3397 for 28 day cycles. Participants will continue to take PLX3397 until disease progression or toxicity.
  Interventions: Drug: PLX3397

INTERVENTIONS:
Drug: PLX3397 — Capsules administered twice daily, continuous dosing. Subjects will take PLX3397 at 1000 mg/day.

SUMMARY:
The main objective of this study is to evaluate the effects of PLX3397 on male subjects with CRPC.

Secondary objectives include evaluating the safety and tolerability of PLX3397 and the anti-tumor effects that PLX3397 has on the the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer, currently with objective progressive disease.
* Castrate level of testosterone (<50 ng/dL).
* Baseline circulating tumor cell (CTC) count ≥10/7.5 mL blood.
* Archival tumor tissue (unstained sections, paraffin block, or frozen tumor tissue) has been requisitioned for shipment to the central laboratory.
* Karnofsky performance status of 80-100.
* Adequate organ and marrow function.

Exclusion Criteria:

* The subject has received:

  * Any systemic chemotherapy (including investigational agents) within 4 weeks (with the exception of nitrosoureas/mitomycin C within 6 weeks), of the first dose of study treatment, OR
  * Biological agents (antibodies, immune modulators, cytokines, or vaccines) within 6 weeks of the first dose of study treatment, OR
  * Hormonal anticancer therapy (not including LHRH agonists or antagonists) within 2 weeks before the first dose of study treatment. Specific restrictions on prior hormonal and other anticancer treatments are detailed in inclusion criterion, OR
  * Small-molecular kinase inhibitors or any other type of investigational agent within 4 weeks before the first dose of study treatment or 5 half-lives of the compound or active metabolite, whichever is shorter.
* The subject has received drugs used to control loss of bone mass (e.g., bisphosphonates) within 4 weeks prior to the first dose of study treatment.
* The subject has symptomatic or uncontrolled brain metastasis or epidural disease requiring current treatment including steroids and anti-convulsants.
* The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) >450 ms at screening.
* The subject has uncontrolled or significant intercurrent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders such as symptomatic congestive heart failure (CHF), *Uncontrolled hypertension
  * Unstable angina pectoris, clinically-significant cardiac arrhythmias
  * History of stroke (including transient ischemic attack [TIA] or other ischemic event) within 6 months of study treatment
  * Myocardial infarction within 6 months of study treatment
  * History of thromboembolic event requiring therapeutic anticoagulation within 6 months of study treatment or main portal vein or vena cava thrombosis or occlusion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-05-25 (Actual); Primary Completion 2013-03-11 (Actual); Study Completion 2013-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6 participants received study drug at 2 clinic sites.
Pre-assignment Details: A total of 20 participants were planned to be enrolled at approximately 2 to 4 clinic sites.
Groups:
- PLX3397: Participants who received a daily oral dose of PLX3397 for 28 day cycles and continued on therapy until disease progression or toxicity.
Period: Overall Study
Arm/Group | PLX3397
Started | 6
Completed | 0
Not Completed | 6
Not completed — Progressive disease (radiographic) | 2
Not completed — Progressive disease (clinical) | 1
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | PLX3397
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (7.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Summary of High Circulating Tumor Cell Count Number In Men With Radiographically Progressive Castration-Resistant Prostate Cancer and High Circulating Tumor Cells
Description: Effects of PLX3397 on CTC number in men with radiographically progressive CRPC and high CTC counts (≥10 CTCs/7.5 mL of blood using CellSearch Assay)
  CTC counts were to be evaluated at the following time points: Screening, Baseline, every 4 weeks after treatment initiation, and at Safety Follow-up.
  Radiographic tumor evaluation were to be performed every 8 weeks. Progression at the first reassessment required a confirmatory scan at a minimum of 6 weeks later, and treatment with study medication was to continue until the progression had been confirmed.
Time Frame: See measure description for time frame.
Population: The study was discontinued and the primary outcome measure was not evaluated. Consequently, no efficacy was evaluated and only safety results are reported. Raw data collected but no efficacy analysis was performed/reported.
Arm/Group | PLX3397
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants Reporting Treatment-Related Adverse Events by System Organ Class and Preferred Term
Time Frame: Assessed from first dose through at least 4 weeks after the last dose.
Population: Adverse events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | PLX3397
Number analyzed (Participants) | 6
Participants
  Anaemia | 1
  Thrombocytopenia | 1
  Constipation | 2
  Diarrhoea | 2
  Nausea | 4
  Fatigue | 3
  Mucosal inflammation | 1
  Alanine aminotransferase increased | 1
  Aspartate aminotransferase increased | 1
  Blood creatinine phosphokinase increased | 1
  Blood glucose increased | 1
  Blood sodium increased | 1
  Lipase increased | 1
  Decreased appetite | 3
  Pain in extremity | 1
  Dyspnoea | 1

3. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events by Worst Severity Grade
Description: Adverse events (AEs) were assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0, where 1=mild, 2=moderate, 3=severe, 4=life-threatening, and 5=death related to AE.
Time Frame: Assessed from first dose through at least 4 weeks after the last dose.
Population: Adverse events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- NCI CTCAE Grade 1: Participants who received PLX3397 and experienced a Grade 1 treatment-emergent adverse event.
- NCI CTCAE Grade 2: Participants who received PLX3397 and experienced a Grade 2 treatment-emergent adverse event.
- NCI CTCAE Grade 3: Participants who received PLX3397 and experienced a Grade 3 treatment-emergent adverse event.
- NCI CTCAE Grade 4: Participants who received PLX3397 and experienced a Grade 4 treatment-emergent adverse event.
- NCI CTCAE Grade 5: Participants who received PLX3397 and experienced a Grade 5 treatment-emergent adverse event.
Arm/Group | NCI CTCAE Grade 1 | NCI CTCAE Grade 2 | NCI CTCAE Grade 3 | NCI CTCAE Grade 4 | NCI CTCAE Grade 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Participants
  Anaemia | 0 | 1 | 0 | 0 | 0
  Thrombocytopenia | 1 | 0 | 0 | 0 | 0
  Constipation | 2 | 0 | 0 | 0 | 0
  Diarrhoea | 2 | 0 | 0 | 0 | 0
  Nausea | 4 | 0 | 0 | 0 | 0
  Fatigue | 1 | 2 | 0 | 0 | 0
  Mucosal inflammation | 1 | 0 | 0 | 0 | 0
  Pyrexia | 0 | 1 | 0 | 0 | 0
  Oedema | 1 | 0 | 0 | 0 | 0
  Oedema peripheral | 1 | 0 | 0 | 0 | 0
  Pain | 2 | 0 | 0 | 0 | 0
  Influenza | 0 | 0 | 1 | 0 | 0
  Pneumonia | 0 | 0 | 1 | 0 | 0
  Fall | 0 | 0 | 1 | 0 | 0
  ALT increased | 0 | 0 | 1 | 0 | 0
  AST increased | 0 | 0 | 1 | 0 | 0
  Blood CPK increased | 0 | 0 | 1 | 0 | 0
  Lipase increased | 0 | 0 | 1 | 0 | 0
  Blood glucose increased | 1 | 0 | 0 | 0 | 0
  Blood sodium increased | 1 | 0 | 0 | 0 | 0
  Decreased appetite | 3 | 0 | 0 | 0 | 0
  Musculoskeletal pain | 1 | 0 | 0 | 0 | 0
  Pain in extremity | 0 | 0 | 1 | 0 | 0
  Peripheral sensory neuropathy | 1 | 0 | 0 | 0 | 0
  Spinal cord disorder | 1 | 0 | 0 | 0 | 0
  Nocturia | 1 | 0 | 0 | 0 | 0
  Urinary retention | 0 | 1 | 0 | 0 | 0
  Pollakiuria | 2 | 0 | 0 | 0 | 0
  Dyspnoea | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from after first dose to 28 days after last dose.
Description: Adverse events that emerge (or worsen) from after the first dose of study drug and within 28 days after last dose.
Arm/Group | PLX3397
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLX3397 (N=6)
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PLX3397 (N=6)
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 3
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatinine phosphokinase increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood sodium increased (Investigations) | 1
Lipase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Spinal cord disorder (Nervous system disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
This study did not meet its planned enrollment goal of 20 participants by the end of 2012. Therefore, enrollment was terminated and efficacy was not evaluated; only the safety results are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No